CLINICAL TRIAL: NCT03368430
Title: Is Dietary Melatonin Supplementation a Viable Adjunctive Therapy for Chronic Periodontitis? A Preliminary Randomized Clinical Trial.
Brief Title: Melatonin as an Adjunctive Therapy for Chronic Periodontitis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hesham El-Sharkawy, Associate Professor of Periodontology and Oral Medicine, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DENT-2017
Record Dates: First submitted 2017-11-29; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Periodontal Diseases
Keywords: Melatonin; Chronic periodontitis; Host modulation therapy
MeSH Terms: conditions — Periodontal Diseases; Chronic Periodontitis | interventions — Melatonin; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | US Export: Yes

ARMS (2):
- Melatonin (Experimental): 10 mg melatonin capsule was given to participants in the test group once per day for only 2 months after performing scaling and root planing (SRP) during the whole 6- month period of the study.
  Interventions: Dietary Supplement: Melatonin
- Placebo (Placebo Comparator): Matching placebo capsule was given to the control group once daily for 2 months after receiving scaling and root planing (SRP) during the whole 6- month period of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — After performing scaling and root planing (SRP) in the test group, melatonin 10 mg oral capsule was taken once daily at night prior to bedtime for only 2 months during the 6-month study period
  Other Names: N-acetyl-5-methoxytryptamine
  Arms: Melatonin
Drug: Placebo — After finishing scaling and root planing (SRP) in the control group, placebo capsule was taken once daily at bedtime for two months.
  Other Names: starch capsule
  Arms: Placebo

SUMMARY:
Background:

Melatonin is an endogenous indoleamine synthesized mainly by pineal gland and showed anti-inflammatory and antioxidant properties. Moreover, melatonin promotes osteoblastic differentiation and suppresses osteoclastic formation. This randomized clinical trial (RCT) was aimed to assess the additive effect of melatonin supplementation in generalized chronic periodontitis (gCP) patients with insomnia who received scaling and root planing (SRP).

Methods:

Seventy four gCP patients with primary insomnia participated in this 6-month RCT and randomly distributed between two groups. Melatonin group (MTN+SRP group, n=38) included patients who were subjected to SRP with a 2- month regimen of 10 mg oral melatonin supplementation capsule once daily at bed-time. In the control group (Placebo+SRP group, n=36), SRP was performed for participants provided with matching placebo capsules. The primary treatment outcome included the clinical attachment gain (CAG) after 3 and 6 months of therapy, whereas, the changes in pocket depth ,bleeding on probing (BOP%) and salivary tumor-necrosis factor-α (TNF-α) levels represented the secondary outcomes.

DETAILED DESCRIPTION:
INTRODUCTION

Chronic periodontitis is a local chronic inflammation of the tooth supporting apparatus initiated by specific microorganisms including Porphyromonas gingivalis, Tannerella forsythia, and Treponema denticola, which are collectively known as the "red complex". It was revealed that periodontal tissue damage begins as inflammatory neutrophil mediated reaction followed by chronic infiltration of monocytes. Previous investigations have reported that most of periodontal tissue destruction is directly caused by the host immune response to the aforementioned specific periodontopathogenic bacteria.

Few years ago, host modulatory therapy (HMT) has emerged as a new concept for the treatment of destructive periodontal diseases. The aim of HMT is to decrease the periodontal tissue damage by reducing the destructive arm of the host immune response and boosting its regenerative features. HMT includes systemically or locally delivered therapeutics which are utilized as adjuncts to conventional periodontal treatment.

A variety of different drugs have been assessed as host modulatory therapeutics such as non-steroidal anti-inflammatory drugs (NSAIDs), tetracyclines and bisphosphonates. Systemic or topical NSAIDs had significant serious adverse events when used for a long time and after stopping their use, a 'rebound' effect' was observed. Subantimicrobial dose of doxycycline (SDD) revealed beneficial outcomes when combined with non surgical treatment of chronic periodontitis; nevertheless, some adverse reactions associated with tetracyclines particularly photosensitivity were noted. Bisphosphonates were proven to significantly increase alveolar bone density and possess anticollgenase activity , however, their long term use could lead to avascular necrosis of jaw bones especially after tooth extraction. Thus, researchers worldwide are continually searching for new host modulatory agents to be used as adjunctive treatments for periodontal disease.

To-date, melatonin (N-acetyl-5-methoxytryptamine) is a well-investigated, endogenous indoleamine which is primarily secreted from the pineal gland and responsible for regulation of sleep/waking cycle. Melatonin possesses a variety of essential properties such as anti-inflammatory, antioxidant, oncostatic and neuroprotective actions. Moreover, melatonin was recently found to promote osteoblastic differentiation and suppress osteoclastic formation through downregulation of the receptor activator of nuclear к-B ligand (RANKL). In lipopolysaccharide-induced experimental periodontitis in rats, locally applied melatonin significantly decreased bone resorption in comparison with rats which received no treatment. Thus, it was proposed that topically applied melatonin can serve as an adjunct to conventional periodontal treatments including scaling and root planing (SRP), as well as, surgical periodontal therapy.

Recent studies have revealed that salivary melatonin levels were significantly reduced in subjects with periodontal disease, suggesting that melatonin could serve as a biomarker for periodontal diagnosis and used as a potential therapeutic in different periodontal diseases. Recently, topical application of 1% melatonin gel on the attached gingivae in diabetic individuals with periodontal disease resulted in significantly decreased pocket depth and gingival index as well as lower levels of serum IL-6 and C-reactive protein after therapy.

Accordingly, we hypothesized that periodontal treatment with daily dietary supplementation of melatonin adjunctive to SRP in generalized chronic periodontitis (gCP) patients suffering from primary insomnia could improve the periodontal outcomes. Hence, the objective of the present clinical trial is to assess whether the adjunctive therapy of daily melatonin supplementation to SRP compared to placebo with SRP, ameliorates clinical periodontal parameters and reduces salivary TNF-α levels after 3 and 6 months of therapy in patients with gCP and primary insomnia.

MATERIALS AND METHODS

Study Population:

The present study was conducted in accordance with the seventh revision of Helsinky declaration in 2013 and approved by the Institutional Review Board (IRB) of Mansoura University. Individuals were selected during their visits to the Periodontics clinics at the Faculty of Dentistry, Mansoura University, from July, 2016 till September , 2017. Individuals were asked to answer prepared questionnaires about their general medical status and sleep/awakening habits followed by diagnosing the periodontal condition to select eligible participants. Patients were considered eligible for participation if they had Athens Insomnia Scale (AIS) score ≥ 6 (provided that individuals have primary insomnia which not related to any other systemic causes or drug intake according to the International Classification of Sleep Disorders , ICSD-3). Each selected patient should have at least 20 teeth. The enrolled patients were diagnosed to have moderate to severe gCP based on Armitage's classification. Exclusion criteria included diabetes mellitus , smokers, individuals having night work shifts, cancer patients , patients with autoimmune diseases or osteoporosis, users of antibiotics or non-steroidal anti-inflammatory drugs within the last 3 months and patients who were subjected to any periodontal therapy during the last year. Enrolled patients signed informed consents prior to their participation in the clinical trial.

Trial design:

Seventy four patients diagnosed with gCP and primary insomnia were randomly assigned by a coin toss to either receive 10 mg oral melatonin capsule (Puritan's Pride, Inc., Holbrook, NY, USA) once per day at bedtime for two months in conjunction with SRP (MTN+SRP group, n = 38), or matching placebo capsules for 2 months plus SRP (Placebo+SRP group, n = 36) in this double-blinded parallel randomized controlled trial (RCT). The randomization process was performed in absence of the working investigators. By a third party (pharmacist), sealed glass bottles were packed with 30 capsules of either melatonin or matching placebo and then coded with specific labels unknown to working investigators and patients. Patients in both groups were instructed to have one capsule at bedtime from the given bottle. Compliance of patients were assessed by counting the left capsules in the returned bottle at the end of each month. Adverse effects of the given drugs were monitored on a weekly basis for two months. All patients received meticulous thorough SRP with an ultrasonic scaler and hand curettes in a single visit by experienced periodontist. For all participants, strict oral hygiene instructions were given and 0.12% chlorhexidine mouthwash was prescribed for two weeks following SRP.

Periodontal records:

Periodontal measures including pocket depth (PD), clinical attachment level (CAL), dichotomous bleeding on probing (BOP) expressed as percentage, gingival (GI) and plaque (PI) indices were recorded at baseline, 3 and 6 months of therapy by a single examiner. To achieve intra-examiner calibration, periodontal mea-surements of 10 patients were performed twice within 2 days prior to RCT conduction. Calibration was approved when measurements of PD and CAL in the two times were within 1 mm variance in more than 90% of all measurements.

Saliva Collection:

Saliva samples were collected in the morning between 8 to 10 a.m. from all participants after fasting overnight. All participants were asked not to have any drinks except water after arousing. Whole unstimulated saliva samples were harvested by expectoration into 5 mL sterile polypropylene tubes before recording the clinical measurements. All saliva samples were centrifuged to remove debris, and immediately frozen and stored at -80οC until evaluation time.

Biochemical Assessment:

TNF-α level was determined in saliva by enzyme-linked immunosorbent assay (ELISA). Saliva samples were pipetted into clean microcap tubes and centrifuged at 10,000 × g for 5 minutes. Then, the supernatants were placed in clean microcap tubes and used immediately for ELISA assay. Human- TNF-α ELISA development kit (R&D systems, Abingdon Science Park,Abingdon, UK) was used to quantify this molecule in saliva samples according to the manufacturers' recommendations. The results of salivary TNF-α assay are expressed as concentrations in nanograms per milliliter.

Trial outcomes:

The primary outcome of the present RCT was the change in clinical attachment gain (CAG) after 3 and 6 months of therapy, whereas, the secondary end-points included the change in pocket depth,BOP% and salivary TNF-α levels after 3 and 6 months.

Assessment of untoward drug effects:

Systemic signs and symptoms were recorded every week after SRP and initiation of medication intake during the first two months. At the end of RCT, patients indicated for additional periodontal treatments were scheduled as necessary.

Statistical Analyses:

This RCT was powered to 80% level to detect an average reduction of PD and CAL equal to 0.5 mm variation between groups. The calculated minimum sample size required to achieve 80% power was 30 patients per group. Kolmogrov-Smirnov test of normality was used to explore data normality. Parametric data were presented as mean ± SD except salivary TNF-α concentrations which were expressed as mean± SEM (standard error of the mean). Baseline data were compared by using Student's t-test. One-way analysis of variance (ANOVA) with Holm-Sidak post hoc correction for multiple comparisons were used to determine significant differences at different time points. The level of significance was adjusted at 5%. Statistical analyses were performed by using the Statistical Package for the Social Sciences v. 20, SPSS, Chi-cago, IL.

ELIGIBILITY:
Inclusion Criteria:

* Patients were considered eligible for participation if they had Athens Insomnia Scale (AIS) score ≥ 6.
* Each selected patient should have at least 20 teeth.
* The enrolled patients were diagnosed to have moderate to severe gCP based on Armitage's classification.

Exclusion Criteria:

* diabetes mellitus.
* smokers.
* individuals having night work shifts.
* cancer patients.
* patients with autoimmune diseases or osteoporosis.
* users of antibiotics or non-steroidal anti-inflammatory drugs within the last 3 months.
* patients who were subjected to any periodontal therapy during the last year.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2016-07-04 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Change of clinical attachment level (clinical attachment gain). | From baseline to 3 and 6 months.
  Clinical attachment level was assessed at baseline,3 and 6 months after receiving scaling and root planing.

SECONDARY OUTCOMES:
Change of pocket depth. | From baseline to 3 and 6 months.
  Pocket depth was measured at baseline,3 and 6 months.
Change of Bleeding on probing. | From baseline to 3 and 6 months.
  Bleeding on probing (0 for absent and 1 for present) was evaluated at baseline and after 3 and 6 months of therapy.
Change of salivary TNF-alpha levels. | From baseline to 3 and 6 months.
  Salivary TNF-alpha levels were measured at baseline and after 3 and 6 months of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hesham M. El-Sharkawy, PhD, Principal Investigator — Mansoura University
Locations (1):
- Faculty of Dentistry, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared after publication of the RCT.

REFERENCES:
- [Background] Wara-aswapati N, Pitiphat W, Chanchaimongkon L, Taweechaisupapong S, Boch JA, Ishikawa I. Red bacterial complex is associated with the severity of chronic periodontitis in a Thai population. Oral Dis. 2009 Jul;15(5):354-9. doi: 10.1111/j.1601-0825.2009.01562.x. Epub 2009 Apr 7. PMID 19371397
- [Background] Lamster IB, Smith QT, Celenti RS, Singer RE, Grbic JT. Development of a risk profile for periodontal disease: microbial and host response factors. J Periodontol. 1994 May;65(5 Suppl):511-20. doi: 10.1902/jop.1994.65.5s.511. PMID 8046567
- [Background] Kantarci A, Van Dyke TE. Lipoxin signaling in neutrophils and their role in periodontal disease. Prostaglandins Leukot Essent Fatty Acids. 2005 Sep-Oct;73(3-4):289-99. doi: 10.1016/j.plefa.2005.05.019. PMID 15979867
- [Background] Page RC. The role of inflammatory mediators in the pathogenesis of periodontal disease. J Periodontal Res. 1991 May;26(3 Pt 2):230-42. doi: 10.1111/j.1600-0765.1991.tb01649.x. PMID 1679130
- [Background] Van Dyke TE, Serhan CN. Resolution of inflammation: a new paradigm for the pathogenesis of periodontal diseases. J Dent Res. 2003 Feb;82(2):82-90. doi: 10.1177/154405910308200202. PMID 12562878
- [Background] Bhatavadekar NB, Williams RC. Modulation of the host inflammatory response in periodontal disease management: exciting new directions. Int Dent J. 2009 Oct;59(5):305-8. PMID 19998666
- [Background] Williams RC. Host modulation for the treatment of periodontal disease. Compend Contin Educ Dent. 2008 Apr;29(3):160-2, 164, 166-8 passim. PMID 18468302
- [Background] Novak MJ, Donley TG. Using host response modifiers in the treatment of periodontal disease. Pract Proced Aesthet Dent. 2002 Nov-Dec;14(9):suppl 3-10; quiz 11. PMID 12685424
- [Background] Krayer JW, Leite RS, Kirkwood KL. Non-surgical chemotherapeutic treatment strategies for the management of periodontal diseases. Dent Clin North Am. 2010 Jan;54(1):13-33. doi: 10.1016/j.cden.2009.08.010. PMID 20103470
- [Background] Moreno Villagrana AP, Gomez Clavel JF. Antimicrobial or subantimicrobial antibiotic therapy as an adjunct to the nonsurgical periodontal treatment: a meta-analysis. ISRN Dent. 2012;2012:581207. doi: 10.5402/2012/581207. Epub 2012 Oct 22. PMID 23150830
- [Background] Rocha ML, Malacara JM, Sanchez-Marin FJ, Vazquez de la Torre CJ, Fajardo ME. Effect of alendronate on periodontal disease in postmenopausal women: a randomized placebo-controlled trial. J Periodontol. 2004 Dec;75(12):1579-85. doi: 10.1902/jop.2004.75.12.1579. PMID 15732857
- [Background] Kos M, Kuebler JF, Luczak K, Engelke W. Bisphosphonate-related osteonecrosis of the jaws: a review of 34 cases and evaluation of risk. J Craniomaxillofac Surg. 2010 Jun;38(4):255-9. doi: 10.1016/j.jcms.2009.06.005. Epub 2009 Jul 9. PMID 19592261
- [Background] Pandi-Perumal SR, BaHammam AS, Brown GM, Spence DW, Bharti VK, Kaur C, Hardeland R, Cardinali DP. Melatonin antioxidative defense: therapeutical implications for aging and neurodegenerative processes. Neurotox Res. 2013 Apr;23(3):267-300. doi: 10.1007/s12640-012-9337-4. Epub 2012 Jun 28. PMID 22739839
- [Background] Joshi N, Biswas J, Nath C, Singh S. Promising Role of Melatonin as Neuroprotectant in Neurodegenerative Pathology. Mol Neurobiol. 2015 Aug;52(1):330-40. doi: 10.1007/s12035-014-8865-8. Epub 2014 Aug 27. PMID 25159482
- [Background] Maria S, Witt-Enderby PA. Melatonin effects on bone: potential use for the prevention and treatment for osteopenia, osteoporosis, and periodontal disease and for use in bone-grafting procedures. J Pineal Res. 2014 Mar;56(2):115-25. doi: 10.1111/jpi.12116. Epub 2014 Jan 15. PMID 24372640
- [Background] Gulle K, Akpolat M, Kurcer Z, Cengiz MI, Baba F, Acikgoz S. Multi-organ injuries caused by lipopolysaccharide-induced periodontal inflammation in rats: role of melatonin. J Periodontal Res. 2014 Dec;49(6):736-41. doi: 10.1111/jre.12156. Epub 2013 Dec 19. PMID 24354339
- [Background] Cutando A, Lopez-Valverde A, de Diego RG, de Vicente J, Reiter R, Fernandez MH, Ferrera MJ. Effect of topical application of melatonin to the gingiva on salivary osteoprotegerin, RANKL and melatonin levels in patients with diabetes and periodontal disease. Odontology. 2014 Jul;102(2):290-6. doi: 10.1007/s10266-013-0122-5. Epub 2013 Aug 11. PMID 23934086
- [Background] Srinath R, Acharya AB, Thakur SL. Salivary and gingival crevicular fluid melatonin in periodontal health and disease. J Periodontol. 2010 Feb;81(2):277-83. doi: 10.1902/jop.2009.090327. PMID 20151807
- [Background] Soldatos CR, Dikeos DG, Paparrigopoulos TJ. The diagnostic validity of the Athens Insomnia Scale. J Psychosom Res. 2003 Sep;55(3):263-7. doi: 10.1016/s0022-3999(02)00604-9. PMID 12932801
- [Background] Ito E, Inoue Y. [The International Classification of Sleep Disorders, third edition. American Academy of Sleep Medicine. Includes bibliographies and index]. Nihon Rinsho. 2015 Jun;73(6):916-23. Japanese. PMID 26065120
- [Background] Armitage GC. Development of a classification system for periodontal diseases and conditions. Ann Periodontol. 1999 Dec;4(1):1-6. doi: 10.1902/annals.1999.4.1.1. PMID 10863370
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464